CLINICAL TRIAL: NCT05829044
Title: Impact of Sex and Age on Non-visual Light Input That Affects Sleep and Circadian Rhythms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth B Klerman MD PhD, Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023P000904
Record Dates: First submitted 2023-04-02; First posted 2023-04-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Normal Physiology
Keywords: eye pupil response; circadian rhythms; light; melatonin

STUDY DESIGN:
Intervention Model Description: All participants will have the same study conditions and schedule except for the order combinations of light stimuli within the pupillometer testing. There are 8 different order combinations of light stimuli. Participants will be randomized to one of those combinations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Testing non-visual light impacts on pupil response, circadian timing, and hormones (Experimental): 1. Pupillometry on day 1 in afternoon and evening and on day 2 in morning and evening. Participants will be randomized to one of 8 different light stimuli within the pupillometry
  2. Red light exposure on night 1 to determine circadian timing
  3. Blue/green light exposure on night 2 to compare hormone response during blue/green light to that during red light on night 1
  Interventions: Device: Pupillometry; Device: Light box exposure

INTERVENTIONS:
Device: Pupillometry — Pupillometer measurement of pupil size in response to different light stimuli
Device: Light box exposure — Using a light box to produce different wavelengths and intensities of light. Exposure to red light on Night 1 and blue/green light on Night 2 to determine circadian timing and suppression of hormone (melatonin)

SUMMARY:
The goal of this clinical trial is to learn how the pupil responds to different light stimuli and how that relates to sleep and daily rhythms in healthy people of different ages.

The main questions it aims to answer are:

* Does the eye's pupil response to light stimuli differ by the sex and age of the participant?
* Is the eye's pupil response to light stimuli related to each participant's sleep timing, their body clock timing, and their hormone responses to light.

Participants will have a special eye exam and complete questionnaires before starting the study to see if they can participate. If they can participate, they will wear a special watch that monitors their activity and light levels for one week. Then they will live in a research room at the Mass General Hospital for 3 days/2 nights during which we will test their pupil response to light, their body clock timing, and their hormone responses to light.

ELIGIBILITY:
Inclusion Criteria:

* (i) 18-85 years old.
* (ii) Habitual sleep onset 10 pm- 1 am (healthy controls only);
* (iii) Habitual wake onset 5:30 am- 8:30 am (healthy controls only);
* (iv) vision correctable to 20/30;
* (v) stable medically.
* (vi) ability to speak, understand, and read English at a high school level

Exclusion Criteria:

* (i) Color blind by Ishihara Color Blindness Test;
* (ii) any history of eye trauma, surgery or abnormality (e.g., retinopathy, glaucoma, cataracts, amblyopia, macular degeneration, congenital color vision deficiencies, or any type of blindness) besides correctable vision abnormalities (e.g., with glasses); any abnormalities on clinical eye exam (e.g., neuritis, Neuromyelitis optica, treated or untreated glaucoma) such that the ophthalmologist recommends the participant not be studied; Limited cataracts (e.g., Lens Opacities Classification (LOCS) III grade <2) will be allowed and documented during the eye exam. Eye drops that affect pupil size or contractility (e.g. mydriatics, miotics); drops to treat glaucoma (e.g., pilocarpine, brimonidine, other drops like artificial tear drops, or anti-inflammatory drops would not be exclusionary)
* (iii) current or history of neurologic or psychiatric disease including autonomic function disorder or migraines; psychiatric disorder requiring medications in a first degree relative (healthy controls only); limited-duration counseling without prescription medications will not be exclusionary; (iv) current or history of circadian rhythm sleep-wake disorder (healthy controls only);
* (v) prescription or non-prescription drugs affecting the pupil (e.g., affecting autonomic function), sleep, melatonin (e.g., lithium, alpha- and beta-adrenergic antagonists), and/or circadian rhythms (e.g., beta blockers, non-steroidal anti-inflammatory drugs, tricyclics);
* (vi) Other disorders that can affect or may be affected by intrinsically photosensitive Retinal Ganglion Cell (ipRGC) function, including diabetes mellitus, multiple sclerosis, Parkinson's disease, seasonal affective disorder;
* (vii) shift- or night-work in past three months; history of night work in preceding 3 year period
* (viii) crossing more than 2 time zones in past three months;
* (ix) presence of depression as assessed by a Beck Depression Inventory (BDI) score >14.
* (x) pregnant or less than 6 weeks post-partum or breast-feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pupil size | During pupillometry testing on Day 1 afternoon, Day 1 evening, Day 2 morning, Day 2 evening
  Pupil size as measured by pupillometry
Melatonin levels for circadian timing assessment | Night 1
  Melatonin levels from saliva collection during Night 1 light box red light exposure
Melatonin levels for hormone response | Night 1 and Night 2
  Melatonin levels from saliva collection during Night 2 light box blue/green light exposure compared to those during Night 1 light box red light exposure

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Klerman, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be conducted per National Institutes of Health (NIH) and MassGeneralBrigham (MGB) policies and regulations. Only de-identified data will be shared.